## Vernon Grant, PhD Assistant Research Professor Center for American Indian and Rural Health Equity Montana State University

NCT05314712

Document date: 01-06-25

## Statistical Analysis Plan

Graphical displays will be used for understanding the data before aggregating and summarizing. For the baseline data, the primary variable of interest is sleep derived from the Pittsburgh Sleep Quality Index survey; sleep will be compared between pre and post intervention using regression approaches with other covariates that have a significant association. It is important to understand the role that these covariates have on sleep. We will also explore other sleep variables that may be indicative of sleep problems. At post intervention (7 weeks), the primary end variable of interest is *change* in sleep (child and adult). Feasibility measures collected at 7-weeks will assess number recruited, number retained, and Blackfoot words, songs, and stories learned.